CLINICAL TRIAL: NCT04066491
Title: A Phase II/III, Multicenter, Randomized, Placebo-controlled Study of Gemcitabine Plus Cisplatin With or Without Bintrafusp Alfa (M7824) as First-line Treatment of Biliary Tract Cancer
Brief Title: Gemcitabine Plus Cisplatin With or Without Bintrafusp Alfa (M7824) in Participants With 1L BTC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Based on a review of data conducted by the Independent Data Monitoring Committee (IDMC), Sponsor decided to discontinue this study as the study was unlikely to achieve the primary objective of overall survival.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200647_0055; 2019-001992-35 (EudraCT Number)
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Results first posted 2022-06-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer
Keywords: Metastatic Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer; Ampullary cancer; M7824; Bintrafusp alfa; Transforming growth factor-beta; Programmed death-ligand 1
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Camurati-Engelmann Syndrome | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-In Part: M7824 + Gemcitabine + Cisplatin (Experimental)
  Interventions: Drug: M7824; Drug: Gemcitabine; Drug: Cisplatin
- Double-blinded Part: M7824 + Gemcitabine + Cisplatin (Experimental)
  Interventions: Drug: M7824; Drug: Gemcitabine; Drug: Cisplatin
- Double-blinded Part: Placebo + Gemcitabine + Cisplatin (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: M7824 — Participants received intravenous infusion of M7824 at a dose of 2400 milligrams (mg), once every 3 weeks (Q3W) 2 years (in case of Complete Response), otherwise until criterion pre-sepcified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 milligram per meter square (mg/m^2) and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks.
  Arms: Double-blinded Part: M7824 + Gemcitabine + Cisplatin; Safety Run-In Part: M7824 + Gemcitabine + Cisplatin
Drug: Placebo — Participants received intravenous infusion of M7824 matched placebo, once every 3 weeks (Q3W) until 2 years (in case of CR), otherwise until crtiterion pre-sepcified in protocol for discontinuation is met.
  Arms: Double-blinded Part: Placebo + Gemcitabine + Cisplatin
Drug: Gemcitabine — Gemcitabine was received intravenously at a dose of 1000 milligram per meter square (mg/m^2) on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks (Q3W).
Drug: Cisplatin — Cisplatin was received intravenously at a dose of 25 mg/m^2 on Day 1 and Day 8 of 21-day cycle, for 8 cycles every 3 weeks (Q3W).

SUMMARY:
Study consisted of an open-label, safety run-in part and a randomized, double-blind, placebo-controlled Phase 2/3 part. In the Phase 2/3 part, the study was evaluated whether bintrafusp alfa in combination with the current standard of care (SoC) (gemcitabine plus cisplatin) improves overall survival (OS) in chemotherapy and immunotherapy-naïve participants with locally advanced or metastatic Biliary Tract Cancer (BTC) compared to placebo, gemcitabine and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Are participants with histologically or cytologically confirmed locally advanced or metastatic BTC
* Participants must have available tumor tissue (primary or metastatic) (archival or fresh biopsies) before the first administration of study treatment
* At least 1 measurable lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 at study entry and at Week 1, Day 1 prior to dosing
* Life expectancy of >= 12 weeks, as judged by the Investigator
* Adequate hematological function, hepatic function, renal function, coagulation function as defined in the protocol
* Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive participants must be treated and on a stable dose of antivirals
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Previous and/or intercurrent cancers
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation, but with the exception of transplants that do not require immunosuppression
* Participants with symptomatic central nervous system (CNS) metastases
* Significant acute or chronic infection including known history of positive test for human immunodeficiency virus (HIV), active tuberculosis, uncontrolled biliary infection and active bacterial or fungal infection requiring systemic therapy (with the exception of hepatitis B and hepatitis C) requiring systemic therapy at study entry and at Week 1 Day 1 prior to dosing.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* History of or concurrent interstitial lung disease
* History of hypersensitivity reactions to bintrafusp alfa, anaphylaxis, or recent (within 5 months) uncontrolled asthma, cardiovascular/cerebrovascular disease
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before randomization
* Prior therapy with any antibody/drug targeting T-cell coregulatory proteins (immune checkpoints)
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (99):
- United States (12):
  - Ironwood Cancer & Research Centers - Chandler II, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Mayo Clinic in Florida - Department of Neurology, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Kansas Medical Center Research Institute, Inc. - University of Kansas Cancer Center/Bloch Pavilion, Westwood, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Methodist Transplant Physicians, Dallas, Texas
  - MD Anderson Cancer Center - Unit 429, Houston, Texas
  - Renovatio Clinical - CENTRAL SITE, The Woodlands, Texas
- Argentina (7):
  - Hospital de Gastroenterologia Dr. Carlos Bonorino Udaondo, Ciudad Autonoma Buenos Aires
  - Instituto de Investigaciones Metabolicas (IDIM), Ciudad Autonoma Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - CEDIT, Salta
  - Centro Medico San Roque S.R.L., San Miguel de Tucumán
  - Fundacion ARS Medica, San Salvador de Jujuy
- Australia (4):
  - Blacktown Hospital - PARENT, Blacktown
  - Monash Health, Clayton
  - Epworth Freemasons, Melbourne
  - Icon Cancer Care South Brisbane, South Brisbane
- Brazil (6):
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos
  - INCA - Instituto Nacional de Câncer, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, Sao Jose Rio Preto
  - A. C. Camargo Cancer Center, São Paulo
  - ICESP - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo
- Chile (5):
  - IC la serena Research, La Serena
  - Centro de Investigación Clínica Bradford Hill, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Prosalud, Santiago
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco
- China (10):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chao Yang Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Hospital, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- France (5):
  - ICO - Site Paul Papin - service d'oncologie medicale, Angers
  - Centre Georges François Leclerc - Oncologie Médicale, Dijon
  - CHU Lille - Hôpital Claude Huriez, Lille
  - ICO - Site René Gauducheau, Saint-Herblain
  - CHU de Toulouse - Hôpital Ranguei, Toulouse
- Germany (5):
  - Vivantes Klinikum Neukoelln - Haematologie und Onkologie, Berlin
  - Universitaetsklinikum Bonn AoeR - Medizinische Klinik I Gastroenterologie, Bonn
  - Universitaetsklinikum Carl Gustav Carus TU Dresden - Medizinische Klinik I, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz - Medizinische Klinik I - HCC Ambulanz, Mainz
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori Milano, Milan
  - IOV - Istituto Oncologico Veneto IRCCS - S.Semplice Dip.Oncologia dei Melanomi, Padua
  - Università Campus Bio-Medico di Roma, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma) - UOC Oncologia, Verona
- Japan (10):
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital - Dept of Hepatobiliary and Pancreatic Oncology, Chūōku
  - NHO Kyushu Cancer Center - Dept of Gastroenterology/Hepatology/Pancreatology, Fukuoka
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of JFCR - Dept of Hepato,Biliary and Pancreatic Medicine, Kōtoku
  - Kyorin University Hospital, Mitaka-shi
  - Aichi Cancer Center Hospital, Nagoya
  - Osaka City University Hospital, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - Kanagawa Cancer Center, Yokohama
- Poland (4):
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Gliwice
  - Pratia, Krakow
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - ETG Zamosc, Zamość
- South Korea (9):
  - Chungnam National University Hospital - Department of Internal Medicine (Rheumatology), Daejeon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Clinic i Provincial de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - Hospital San Pedro de Alcantara - Servicio de Oncologia, Cáceres
  - Hospital Universitario Reina Sofia - Dept of Oncology, Córdoba
  - ICO l´Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital Universitario Clinico San Carlos - Servicio de Oncologia, Madrid
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia - Servicio de Hematologia y Oncologia Medica, Valencia
  - Hospital Universitari i Politecnic La Fe - Servicio de Oncologia Medica, Valencia
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- The Christie - Dept of Oncology, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union.
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Yoo C, Oh DY, Choi HJ, Kudo M, Ueno M, Kondo S, Chen LT, Osada M, Helwig C, Dussault I, Ikeda M. Phase I study of bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1, in patients with pretreated biliary tract cancer. J Immunother Cancer. 2020 May;8(1):e000564. doi: 10.1136/jitc-2020-000564. PMID 32461347
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0055
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 2 parts: Safety run-in part and double-blind part. Participants who enrolled in safety run-in part of study were not eligible to participate in double-blind part.
Groups:
- Safety Run-In Part: M7824 + Gemcitabine + Cisplatin: Participants received intravenous infusion of M7824 at a dose of 2400 milligrams (mg), once every 3 weeks (Q3W) 2 years (in case of Complete Response), otherwise until criterion pre-specified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 milligram per meter square (mg/m^2) and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks.
- Double-blinded Part: Placebo + Gemcitabine + Cisplatin: Participants received intravenous infusion of M7824 matched placebo, once every 3 weeks (Q3W) until 2 years (in case of CR), otherwise until crtiterion pre-sepcified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 mg/m^2 and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks. In case of any missed dose for chemotherapy, gemcitabine and cisplatin combination administered on Day 15 of that cycle or at the end of the scheduled 8 cycles (up to 16 administrations of gemcitabine and cisplatin combination). The administration of the missed dose on Day 15 or at the end of 8 cycles is Investigator's clinical decision.
- Double-blinded Part: M7824 + Gemcitabine + Cisplatin: Participants received intravenous infusion of M7824 at a dose of 2400 milligrams (mg), once every 3 weeks (Q3W) 2 years (in case of CR), otherwise until crtiterion pre-sepcified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 mg/m^2 and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks. In case of any missed dose for chemotherapy, gemcitabine and cisplatin combination administered on Day 15 of that cycle or at the end of the scheduled 8 cycles (up to 16 administrations of gemcitabine and cisplatin combination). The administration of the missed dose on Day 15 or at the end of 8 cycles is Investigator's clinical decision.
Period: Overall Study
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Started | 12 | 149 | 148
Treated | 12 | 149 | 146
Completed | 12 | 149 | 146
Not Completed | 0 | 0 | 2
Not completed — Randomized, not treated | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin | Total
Number analyzed (Participants) | 12 | 149 | 148 | 309
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (11.9) | 64 (10.6) | 63 (10.8) | 63 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 78 | 68 | 151
  Male | 7 | 71 | 80 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 21 | 22 | 44
  Not Hispanic or Latino | 11 | 128 | 126 | 265
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 6 | 93 | 90 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 51 | 51 | 108
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in Part: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: A DLT is a toxicity related to the study intervention that meets the following criteria as evaluated in the open-label, safety run-in: Grade 3 or 4 Immune-related adverse event (irAE) that needs permanent discontinuation of M7824 treatment; a malignant skin lesion induced by M7824 that is local and can be resected with a negative resection margin is not a DLT; Grade 3 or 4 nonhematologic toxicity other than irAE, A life threatening hematological toxicity (unless clearly attributable to chemotherapy alone), which is hardly medically manageable, including a bleeding event resulting in urgent intervention and admission to an intensive care unit and Grade 5 toxicity.
Time Frame: Day 1 up to Day 21 of Cycle 1 (each Cycle is of 21 days)
Population: The DLT analysis set included all participants who experienced at least one DLT (either by Investigator or by Safety Monitoring Committee (SMC) or who completed the safety run-in, that is the 21-day DLT evaluation period, receiving at least one infusion of M7824 and of both gemcitabine and cisplatin and not being withdrawn during the DLT evaluation period for reasons other than toxicity.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-In Part: M7824 + Gemcitabine + Cisplatin: Participants received intravenous infusion of M7824 at a dose of 2400 milligrams (mg), once every 3 weeks (Q3W) 2 years (in case of Complete Response), otherwise until criterion pre-specified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 mg/m^2 and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks.
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Double-blind Part: Overall Survival
Description: Overall Survival was defined as the time from study day 1 to the date of death due to any cause. The overall survival was analyzed by using the Kaplan-Meier method.
Time Frame: Time from study day 1 up to data cutoff (assessed up to 609 days)
Population: Intent-to-Treat analysis set included all randomized participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 18 | 23
Months | 11.5 [0.9 to 15.2] | 11.5 [0.2 to 13.9]

3. Secondary Outcome: Safety Run-in Part: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs) and Treatment Related TEAEs According to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE was defined as events with onset date or worsening during the on treatment period. TEAEs included serious TEAEs and non-serious TEAEs.
Time Frame: Time from first treatment up to data cutoff (assessed up to 609 days)
Population: The safety run-in (SRI) analysis set includes all participants from the safety run-in part who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 12
Participants
  Participants with TEAEs | 12
  Participants with Serious TEAEs | 5
  Participants with Treatment-related TEAEs | 11

4. Secondary Outcome: Safety Run-in Part: Number of Participants With Grade Greater Than or Equal (>=) 3 Laboratory Abnormalities
Description: Laboratory investigation included hematology and biochemistry. The number of participants with Grade >=3 laboratory abnormalities were reported. Severity of grade 3 or higher TEAEs were graded using NCI-CTCAE v5.0 toxicity grades, as follows: Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: Time from first treatment up to data cutoff (assessed up to 609 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-In Part: M7824 + Gemcitabine + Cisplatin: Participants received intravenous infusion of M7824 at a dose of 2400 milligrams (mg), once every 3 weeks (Q3W) 2 years (in case of Complete Response), otherwise until criterion pre-specified in protocol for discontinuation is met, in combination with intravenous infusion of Gemcitabine and Cisplatin at a dose of 1000 mg/m^2 and 25 mg/m^2 respectively on Day 1 and Day 8 of 21- day cycle, for 8 cycles every 3 weeks. In case of any missed dose for chemotherapy, gemcitabine and cisplatin combination administered on Day 15 of that cycle or at the end of the scheduled 8 cycles (up to 16 administrations of gemcitabine and cisplatin combination). The administration of the missed dose on Day 15 or at the end of 8 cycles is Investigator's clinical decision.
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 12
Participants
  Hemoglobin low | 6
  Leukocytes low | 4
  Neutrophils low | 6
  Platelets low | 3
  Alanine Aminotransferase high | 2
  Bilirubin high | 1
  Creatinine high | 1
  Lipase high | 1
  Potassium low | 1
  Lymphocytes low | 2
  Corrected Calcium high | 1

5. Secondary Outcome: Double-blind Part: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Independent Review Committee (IRC)
Description: Progression free survival was defined as the time from randomization of study intervention until the first documentation of disease progression (PD) or death due to any cause in the absence of documented PD, whichever occurred first. PD: At least a 20 percent (%) increase in the sum of the longest diameter (SLD) taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from randomization of study drug until the first documentation of PD or death, assessed up to 609 days
Population: The intent-to-treat (ITT) analysis set includes all randomized participants. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 44 | 49
Months | 5.6 [4.2 to 6.9] | 5.5 [2.8 to 6.7]

6. Secondary Outcome: Double-blind Part: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: Percentage of participants with confirmed objective response that is at least one overall assessment of complete response (CR) or partial response (PR) reported here. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by IRC.
Time Frame: Time from randomization of study drug up to data cut off (assessed up to 609 days)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 77 | 73
Percentage of participants | 19.5 [11.3 to 30.1] | 31.5 [21.1 to 43.4]

7. Secondary Outcome: Double-blind Part: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: DOR was defined for participants with objective response, as the time from first documentation of objective response (confirmed Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC. Results were calculated based on Kaplan-Meier estimates.
Time Frame: From first documented objective response to PD or death due to any cause, assessed up to 609 days
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 7 | 9
Months | 12.5 [2.7 to 12.5] | 7.0 [1.4 to 8.3]

8. Secondary Outcome: Double-blind Part: Durable Response of at Least 6 Months According to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 as Assessed by Investigator
Description: Durable Response was defined as the number of participants with confirmed objective response (CR or PR) according to RECIST 1.1, determined by Investigator with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions.
Time Frame: Time from first treatment assessed up to 1148 days
Population: Based on a review of data conducted by the Independent Data Monitoring Committee (IDMC), Sponsor decided to discontinue this study as the study was unlikely to achieve the primary objective of overall survival. Subsequently, the data for this outcome measure was not collected and analyzed.
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Double-blind Part: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (SAEs), Treatment Related TEAEs and Adverse Events of Special Interest (AESIs) According to NCI-CTCAE Version 5.0
Description: AE was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAE was defined as events with onset date or worsening during the on treatment period. TEAEs included serious TEAEs and non-serious TEAEs. Adverse events of special interest (AESI) are serious or non-serious AEs that are of clinical interest and should be closely followed. For this study, AESIs include the following: Infusion-related reactions including immediate hypersensitivity; Immune-related AEs; Transforming growth factor beta (TGFβ) inhibition mediated skin reactions; Anemia; Bleeding AEs.
Time Frame: Time from first treatment up to data cutoff (assessed up to 609 days)
Population: Safety analysis set included all participants who were administered at least one dose of any study treatment (M7824, placebo, gemcitabine or cisplatin).
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
Number analyzed (Participants) | 149 | 146
Participants
  Participants with TEAEs | 145 | 140
  Participants with Serious TEAEs | 36 | 58
  Participants with Treatment-related TEAEs | 136 | 133
  Participants with AESIs | 8 | 16

ADVERSE EVENTS:
Time Frame: Time from first treatment up to data cutoff (assessed up to 609 days)
Description: Safety Run-In Part: The safety run-in (SRI) analysis set includes all participants from the safety run-in part who were administered any dose of any study intervention and double-blinded part safety analysis set included all randomized participants who were administered at least one dose of study treatment (M7824, Placebo, Gemcitabine or Cisplatin).
Arm/Group | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin | Double-blinded Part: Placebo + Gemcitabine + Cisplatin | Double-blinded Part: M7824 + Gemcitabine + Cisplatin
All-Cause Mortality (participants affected / at risk) | 7/12 | 26/149 | 31/146
Serious Adverse Events (participants affected / at risk) | 5/12 | 36/149 | 58/146
Other Adverse Events (participants affected / at risk) | 12/12 | 142/149 | 134/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin (N=12) | Double-blinded Part: Placebo + Gemcitabine + Cisplatin (N=149) | Double-blinded Part: M7824 + Gemcitabine + Cisplatin (N=146)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 4
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 3 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 5 | 6
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 2
Biliary sepsis (Infections and infestations) | 0 | 0 | 2
Biliary tract infection (Infections and infestations) | 0 | 3 | 2
COVID-19 (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Herpes simplex encephalitis (Infections and infestations) | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 3 | 2
Blood sodium decreased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 2 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Device occlusion (Product Issues) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-In Part: M7824 + Gemcitabine + Cisplatin (N=12) | Double-blinded Part: Placebo + Gemcitabine + Cisplatin (N=149) | Double-blinded Part: M7824 + Gemcitabine + Cisplatin (N=146)
Anaemia (Blood and lymphatic system disorders) | 6 | 79 | 78
Leukopenia (Blood and lymphatic system disorders) | 1 | 7 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 40 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 12 | 14
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 3
Eye pain (Eye disorders) | 1 | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 11 | 13
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 5
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 9 | 1
Constipation (Gastrointestinal disorders) | 4 | 51 | 40
Diarrhoea (Gastrointestinal disorders) | 3 | 15 | 20
Dyspepsia (Gastrointestinal disorders) | 1 | 10 | 6
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 13
Nausea (Gastrointestinal disorders) | 6 | 72 | 64
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 6 | 16
Vomiting (Gastrointestinal disorders) | 1 | 32 | 31
Asthenia (General disorders) | 2 | 18 | 23
Fatigue (General disorders) | 4 | 35 | 29
Generalised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 11 | 5
Mucosal inflammation (General disorders) | 1 | 4 | 1
Oedema peripheral (General disorders) | 1 | 10 | 9
Pyrexia (General disorders) | 3 | 19 | 33
Cholangitis (Hepatobiliary disorders) | 1 | 3 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 4
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 4 | 9
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 6
Alanine aminotransferase increased (Investigations) | 2 | 20 | 13
Amylase increased (Investigations) | 2 | 8 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 22 | 13
Blood albumin decreased (Investigations) | 1 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 8 | 7
Blood bilirubin increased (Investigations) | 0 | 14 | 9
Blood creatinine increased (Investigations) | 1 | 7 | 6
Blood magnesium decreased (Investigations) | 1 | 3 | 2
Creatinine renal clearance decreased (Investigations) | 1 | 9 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 10 | 4
Haemoglobin decreased (Investigations) | 1 | 0 | 3
Iron binding capacity total decreased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 9 | 5
Neutrophil count decreased (Investigations) | 5 | 59 | 28
Platelet count decreased (Investigations) | 3 | 38 | 34
White blood cell count decreased (Investigations) | 3 | 36 | 19
Decreased appetite (Metabolism and nutrition disorders) | 3 | 36 | 30
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 10 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 13 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 8 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 10 | 0
Dizziness (Nervous system disorders) | 0 | 13 | 8
Dysgeusia (Nervous system disorders) | 2 | 3 | 6
Headache (Nervous system disorders) | 0 | 13 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 5
Taste disorder (Nervous system disorders) | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 6 | 3
Insomnia (Psychiatric disorders) | 1 | 2 | 12
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 19
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 16 | 5
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 14 | 35
Rash (Skin and subcutaneous tissue disorders) | 6 | 21 | 36
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4 | 10
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 6 | 3
Hypertension (Vascular disorders) | 1 | 11 | 6

LIMITATIONS AND CAVEATS:
Data collection and analysis of Pharmacokinetics and Immunogenicity were omitted and not conducted due to business reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT04066491/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT04066491/SAP_001.pdf